CLINICAL TRIAL: NCT01759602
Title: Phase 1b Study of C1-esterase Inhibitor (Cinryze) With Standard of Care for Acute Treatment of Neuromyelitis Optica Exacerbations
Brief Title: C1-esterase Inhibitor (Cinryze) for Acute Treatment of Neuromyelitis Optica Exacerbation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Levy (Other)
Collaborators: ViroPharma (Industry)
Responsible Party: Sponsor-Investigator, Michael Levy, Assistant Professor, Johns Hopkins University
Organization: Johns Hopkins University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00078437
Record Dates: First submitted 2012-12-29; First posted 2013-01-03 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Neuromyelitis Optica
Keywords: Neuromyelitis optica; Devic's disease; NMO; Devic
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Complement C1 Inhibitor Protein; SERPING1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- C1-esterase inhibitor (Cinryze) (Experimental): This is a phase 1b open-label, interventional proof-of-concept study in patients with neuromyelitis optica (NMO) in which all subjects will receive 3 daily infusions of 2000 Units of intravenous CINRYZE at the onset of an NMO exacerbation in addition to standard of care high-dose steroids, plus an additional 2 infusions of 1000 Units of intravenous CINRYZE during a second treatment phase with plasma exchange, if necessary.
  Interventions: Drug: C1-esterase inhibitor (Cinryze)

INTERVENTIONS:
Drug: C1-esterase inhibitor (Cinryze)
  Other Names: Cinryze

SUMMARY:
The overall objective is to evaluate the tolerability/safety and preliminary efficacy of CINRYZE® (C1 esterase inhibitor [human]) as add-on therapy for treatment of acute optic neuritis and/or transverse myelitis in NMO and NMOSD.

Primary Objective: To evaluate the safety and tolerability of 3-5 doses of 1000 - 2000 Units intravenous CINRYZE in NMO/NMOSD patients during an acute exacerbation.

Secondary Objectives:

* To determine the frequency of adverse events with CINRYZE in this patient population.
* To determine the effect of CINRYZE on NMO clinical scores (Expanded Disability Status Scale and Low Contrast Visual Acuity).
* To compare the change in MRI lesion size and extent following a course of CINRYZE.

DETAILED DESCRIPTION:
The rationale for using C1-esterase inhibitor (CINRYZE) in NMO is based on pathology showing a role for complement in active NMO lesions. NMO is not unique in involving complement, which may have a pathogenic role in other demyelinating diseases including multiple sclerosis. However, NMO is characterized by its complement involvement depositing in a rim or rosette pattern in all/most active lesions. In vitro, complement mediates damage initiated by anti-AQP4 antibody binding to astrocytes. The effector of antibody triggered cell damage is the complement cascade and blocking the complement cascade with C1-inhibitor prevents damage ex vivo. Based on mounting evidence, the consensus in the field is that prevention of the complement cascade in the CNS would ameliorate the damage caused in NMO inflammatory attacks. In contrast to a prevention trial, this study would provide for complement inhibition only during an active NMO attack. This approach is designed to administer the inhibitory drug when complement damage is at its peak which minimizes adverse effects from prolonged complement inhibition.

Patients with NMO do not lack natural C1-esterase inhibitor, but artificially tipping the balance to suppress the complement pathways using purified human C1-esterase inhibitor in patients with hyperactive complement activation has been shown to be beneficial in myocardial infarction and sepsis. Similarly, the rationale for adding human C1-esterase inhibitor to the treatment for NMO acute exacerbations is to tip the balance toward complement suppression in an effort to reduce complement-mediated neurologic damage.

This is a phase 1b open-label, interventional proof-of-concept study in which all subjects will receive 3 daily infusions of 2000 Units of intravenous CINRYZE at the onset of an NMO exacerbation, plus an additional 2 infusions of 1000 Units of intravenous CINRYZE during a second treatment phase with plasma exchange, if necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent.
2. 18-65 years of age.
3. New acute optic neuritis and/or transverse myelitis. A clinical event is defined as an episode of inflammation in the spinal cord and/or optic nerve leading to neurologic symptoms not ascribed to another disease process.
4. Diagnosis of NMO according to the 2006 revisions of the Wingerchuk diagnostic criteria for NMO (Wingerchuk, 2006), or AQP4 positive NMOSD per the EFNS Guidelines. For NMO, subjects must have two absolute criteria:

   1. optic neuritis
   2. myelitis and at least two of three supportive criteria:
   3. presence of a contiguous spinal cord MRI lesion extending over three or more vertebral segments,
   4. MRI criteria NOT satisfying the revised McDonald diagnostic criteria for MS [Polman, 2011]
   5. NMO-IgG (AQP4) in serum. For NMOSD, subjects must have longitudinally extensive transverse myelitis (LETM) recurrent isolated optic neuritis (RION)/bilateral optic neuritis (BON), or opticospinal multiple sclerosis (OSMS) that is AQP4 antibody positive.
5. A female subject is eligible to enter the study if she is:

A. Not pregnant or nursing; B. Of non-childbearing potential (i.e. women who have had a hysterectomy, are post-menopausal, which is defined as >2 years without menses or, in female subjects who have been post-menopausal for <2 years, must be confirmed with Follicle Stimulating Hormone (FSH) and estradiol levels), have both ovaries surgically removed or have current documented tubal ligation) OR Of child-bearing potential (i.e. women with functional ovaries and no documented impairment of oviductal or uterine function that would cause sterility). This category includes women with oligomenorrhoea (even severe), women who are perimenopausal or have just begun to menstruate.

C. Subject has a negative serum pregnancy test at screening and agrees to one of the following:

1. Complete abstinence from intercourse for the period from consent into the study until 6 months after the last dose of investigational product; or,
2. Consistent and correct use of one of the following acceptable methods of birth control for the period from consent into the study until 6 months after the last dose of investigational product:

i. Oral contraceptives (either combined or progesterone only) ii. Injectable progesterone iii. Levonorgestrel implants iv. Estrogenic vaginal ring v. Percutaneous contraceptive patches vi. Intrauterine device (IUD) or intrauterine system (IUS) with a documented failurerate of <1% per year vii. Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study; this male must be the sole partner for the subject viii. Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository).

Exclusion Criteria:

1. Current evidence or known history of clinically significant infection including:

   1. Chronic or ongoing active infectious disease requiring long term systemic treatment such as, but not limited to: PML, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis, or active hepatitis C.
   2. Previous serious opportunistic or atypical infections.
   3. History of positive serology for hepatitis B.
   4. Prior history, or suspicion, of tuberculosis (TB)
   5. History of positive serology for HIV.
2. History of clinically significant CNS trauma (e.g. traumatic brain injury, cerebral contusion, spinal cord compression).
3. History or presence of myelopathy due to spinal cord compression by disc or vertebral disease.
4. Past or current history of medically significant adverse effects (including allergic reactions) from:

   a. Corticosteroids
5. Past or current malignancy, except for

   1. Cervical carcinoma Stage 1B or less
   2. Non-invasive basal cell and squamous cell skin carcinoma
   3. Cancer diagnoses with a duration of complete response (remission) >5 years
   4. A history of hematologic malignancy excludes a subject from participation, regardless of response.
6. Significant concurrent, uncontrolled medical condition including, but not limited to, cardiac, renal, hepatic, hematological, gastrointestinal, endocrine, immunodeficiency syndrome, pulmonary, cerebral, psychiatric, or neurological disease which could affect the subject's safety, impair the subject's reliable participation in the trial, impair the evaluation of endpoints, or necessitate the use of medication not allowed by the protocol, as determined by the PI of the study.
7. Use of an investigational drug or other experimental therapy for a condition other than NMO within 4 weeks, 5 pharmacokinetic half lives or duration of biological effect (whichever is longer) prior to screening.
8. Current participation in any other interventional clinical trial. Participation in non-interventional trial requires approval of the protocol by investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levy, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Tradtrantip L, Asavapanumas N, Phuan PW, Verkman AS. Potential therapeutic benefit of C1-esterase inhibitor in neuromyelitis optica evaluated in vitro and in an experimental rat model. PLoS One. 2014 Sep 5;9(9):e106824. doi: 10.1371/journal.pone.0106824. eCollection 2014. PMID 25191939
- See also: Johns Hopkins NMO Research Lab — http://www.hopkinsmedicine.org/neurology_neurosurgery/research/neuromyelitis-optica-research-lab/

RESULTS

PARTICIPANT FLOW:
Groups:
- C1-esterase Inhibitor (Cinryze): This is a phase 1b open-label, interventional proof-of-concept study in patients with neuromyelitis optica (NMO) in which all subjects will receive 3 daily infusions of 2000 Units of intravenous CINRYZE at the onset of an NMO exacerbation in addition to standard of care high-dose steroids, plus an additional 2 infusions of 1000 Units of intravenous CINRYZE during a second treatment phase with plasma exchange, if necessary.
  C1-esterase inhibitor (Cinryze)
Period: Overall Study
Arm/Group | C1-esterase Inhibitor (Cinryze)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | C1-esterase Inhibitor (Cinryze)
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 41 [21 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Safety Events During Hospitalization
Description: Over the course of hospitalization for the acute NMO exacerbations, subjects will be monitored daily for frequency of adverse events.
Time Frame: 5-21 days
Measure: Number; unit: adverse safety events
Arm/Group | C1-esterase Inhibitor (Cinryze)
Number analyzed (Participants) | 10
adverse safety events | 0

2. Secondary Outcome: Frequency of Serious Adverse Events.
Time Frame: 5-21 days
Measure: Number; unit: serious adverse events
Arm/Group | C1-esterase Inhibitor (Cinryze)
Number analyzed (Participants) | 10
serious adverse events | 0

3. Secondary Outcome: Percentage of Subjects Withdrawing Due to Adverse Events.
Time Frame: 5-21 days
Measure: Number; unit: percentage of subjects withdrawing
Arm/Group | C1-esterase Inhibitor (Cinryze)
Number analyzed (Participants) | 10
percentage of subjects withdrawing | 0

4. Secondary Outcome: Change From Baseline in Hematology, Chemistry, and Urinalysis Parameters.
Description: ALT elevations were considered "mild" if they rose to less than 4-fold baseline levels.
Time Frame: 5-21 days
Measure: Number; unit: participants
Arm/Group | C1-esterase Inhibitor (Cinryze)
Number analyzed (Participants) | 10
participants
  ALT Level, mild elevation | 1
  Hematology, abnormal | 0
  Urinalysis, abnormal | 0

5. Secondary Outcome: Expanded Disability Status Score (EDSS)
Description: The Kurtzke Expanded Disability Status Scale (EDSS) was developed to measure the disability status of patients with multiple sclerosis. It allows an objective quantification of the level of functioning that could be widely and reproducibly used by researchers and health care providers.
  The EDSS provides a total score on a scale that ranges from 0 to 10. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refer to the loss of ambulatory ability. The range of main categories include (0) = normal neurologic exam; to (5) = ambulatory without aid or rest for 200 meters; disability severe enough to impair full daily activities; to (10) = death due to MS. In addition, it also provides eight subscale measurements called Functional System (FS) scores.
Time Frame: participants were followed for the duration of hospital stay ranging from 5-21 days, an average of 13 days; EDSS assessment was administered at discharge
Measure: Median (Full Range); unit: EDSS scores
Arm/Group | C1-esterase Inhibitor (Cinryze)
Number analyzed (Participants) | 10
EDSS scores | 2.5 [0 to 8]

ADVERSE EVENTS:
Arm/Group | C1-esterase Inhibitor (Cinryze)
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No